CLINICAL TRIAL: NCT06615076
Title: Enhancing Care and Outcomes for Patients with Hypertensive Disorders of Pregnancy and Diabetes During the First Postpartum Year: a Randomized Control Trial
Brief Title: Enhancing Care & Outcomes for Patients During the First Postpartum Year
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Jenifer Fahey, Principal Investigator, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HP-00107491
Record Dates: First submitted 2024-09-12; First posted 2024-09-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Postpartum Period; Pregnancy; Hypertension, Pregnancy Induced
MeSH Terms: conditions — Hypertension, Pregnancy-Induced

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The intervention group will have scheduled structured postpartum visits at 3, 6, and 12 months with obstetric care providers. These structured visits will be targeted at both managing current hypertensive and/or diabetes disorders and decreasing the risk of developing these disorders. Additional postpartum and primary care concerns will also be addressed as they arise.
  Interventions: Other: Postpartum Visits
- Control (Active Comparator): The control group will have study assessment visits at 3, 6, and 12 months during the first postpartum year, conducted by a Registered Nurse (RN).
  Interventions: Other: Postpartum Visits

INTERVENTIONS:
Other: Postpartum Visits — Postpartum visits with obstetric care providers
  Arms: Intervention
Other: Postpartum Visits — Postpartum visits with study RN.
  Arms: Control

SUMMARY:
The United States is in the midst of a maternal mortality and morbidity crisis, with more than half of maternal deaths occurring within the first postpartum year. Patients with hypertensive disorders of pregnancy (HDP) and diabetes have been found to be particularly high-risk, as they have a significantly increased risk for the development of cardiovascular disease in the long-term postpartum period. Traditionally, postpartum care has consisted of a single office visit at six weeks postpartum. Recent research has suggested that postpartum care should be an ongoing process, tailored to each woman's specifics needs. The purpose of this research study is to evaluate the effectiveness of obstetric care providers as primary care providers for patients at increased risk of maternal morbidity and mortality in the full first postpartum year.

DETAILED DESCRIPTION:
Maternal mortality rates (MMR) and rates of pregnancy-related deaths continue to worsen in the United States (U.S.), with more women dying per capita as a result of complications from pregnancy and childbirth than in any other high-income nation. Persistent and stark racial disparities exist in U.S. rates of maternal deaths and severe maternal morbidity, with Black women being 2.6 times more likely to die than White women. The Centers for Disease Control & Prevention (CDC) estimate that 69% of pregnancy-related deaths occur within the postpartum period, with 36% occurring up to one week after delivery and 33% occurring up to one year after delivery. It is estimated that 60% of maternal deaths are preventable. This fact, along with the rise in postpartum maternal mortality suggests there are unmet medical needs during this time interval.

Hypertensive disorders in pregnancy (HDP), defined as pre-pregnancy (chronic) or pregnancy-associated hypertension, are the most common complication observed during pregnancy, affecting 8%-10% of all pregnancies in the United States. HDP continue to be among the leading causes of pregnancy-related maternal mortality worldwide and contribute to 7% of pregnancy-related maternal deaths in the United States annually. Additionally, the rates of HDP align with the racial disparities seen in maternal morbidity and mortality, with Black and American Indian and Alaska Native women being affected two to three times more than non-Hispanic White women. Despite being a leading cause of severe maternal morbidity and mortality during pregnancy and in the postpartum period, HDPs are preventable. Close monitoring of BP and timely intervention are essential for reducing morbidity in women with HDP, especially preeclampsia, due to the progressive nature of the disease. The American College of Obstetricians and Gynecologists (ACOG) recommends BP monitoring throughout pregnancy, as well as at 72-hour postpartum and again between 7-10 days postpartum.

The prevalence of gestational diabetes, which is the onset of glucose intolerance within pregnancy, has steadily risen in the United States, increasing from 6.0% in 2016 to 8.3% in 2021. Gestational diabetes has become an indicator of future cardiovascular disease and an established threat of maternal morbidity and mortality. Accordingly, the American College of Obstetricians and Gynecologists (ACOG) and the American Diabetes Association (ADA) stress the importance of screening women with a prior diagnosis of gestational diabetes for continued glucose intolerance at six weeks postpartum and at least once every 3 years after pregnancy.

ACOG states that the weeks following birth are a critical period for a woman and her infant, setting the stage for long-term health outcomes and well-being. ACOG recommends postpartum care should be an ongoing process rather than a single encounter to optimize the health of women and infants. Postpartum follow-up beyond the traditional 6-week visit is particularly important for women with medical complications during pregnancy. Lack of insurance and lack of primary care provider have been cited as obstacles to this follow-up in low-income individuals. Research suggests that obstetric care providers can be effective PCPs and that many patients of reproductive age consider and prefer their obstetric or gynecologic care provider to be their PCP and may not visit another PCP regularly.

The Maryland legislature recently passed Senate Bill 923 which requires Medicaid to extend postpartum coverage for eligible pregnant women from 2 months to 12 months immediately following the end of the women's pregnancy. Postpartum coverage changes began April 1, 2022. Maryland is nationally on the forefront of this initiative, with few other states having enacted this legislation previously. The University of Maryland Medical System is uniquely poised and obligated, as Maryland's state hospital and hospital network, to enact proactive workflows and interventions to take advantage of this Medicaid expansion to improve patient care and outcomes for patients who develop hypertensive disorders of pregnancy during the first year postpartum. Patients of color and patients who receive Medicaid are disproportionately at risk for HDP and diabetes, are a large part of the systems patient population, and could benefit from increased longitudinal care with their OB providers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Pregnant individuals
* Planning to deliver and continue postpartum care at the University of Maryland Medical Center
* Diagnosis of HDP or diabetes (pre-gestational or gestational) before discharge from admission for delivery
* Medicaid insurance coverage

Exclusion Criteria:

* Less than 18 years of age
* Fetal demise
* No diagnosis of HDP and/or diabetes (pre-gestational or gestational)
* Non-Medicaid insurance coverage

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in systolic blood pressure measurement from baseline | 6 weeks, 3, 6, and 12 months postpartum
  Diagnosis and treatment of hypertension through systolic blood pressure measurement by 12 months postpartum. An increase in systolic blood pressure would indicate continued and/or worsening hypertension.
Change in diastolic blood pressure measurement form baseline | 6 weeks, 3, 6, and 12 months postpartum
  Diagnosis and treatment of hypertension through diastolic blood pressure measurement by 12 months postpartum. An increase in diastolic blood pressure would indicate continued and/or worsening hypertension.
Change from baseline in blood glucose level measured by fingerstick | 6 weeks, 3, 6, and 12 months postpartum
  Diagnosis and treatment of diabetes through blood glucose measurement by fingerstick by 12 months postpartum. An increase from baseline in blood glucose would indicate diabetes.
Change in serum A1C level from baseline | 6 and 12 months postpartum
  Diagnosis and treatment of diabetes through serum A1C measurement by 12 months postpartum. An increase in A1C levels would indicate pre-diabetes or diabetes.

SECONDARY OUTCOMES:
Postpartum depression severity assessed using Edinburgh Depression Scale (EPDS) | 6 weeks and 3, 6, and 12 months postpartum
  Patient screening using the Edinburgh Perinatal Depression Scale (EPDS), which is a 10-item validated scale that measures depressive symptoms and is designed for use with pregnant and postpartum women. Each question has four ordinal response options, which can give a total score from 0 to 30, with higher scores indicating more severe symptoms.
Postpartum anxiety severity assessed using Generalized Anxiety Disorder Questionnaire (GAD-7) | 6 weeks and 3, 6, and 12 months postpartum
  Patient screening using the Generalized Anxiety Disorder Questionnaire (GAD-7), a 7-item validated scale used to screen for symptoms of anxiety. The questions can yield a total score between 0-21, with higher scores indicating more severe symptoms.
Change in weight measured by change in kilograms from baseline | 3, 6, and 12 months postpartum
  Measurement of postpartum weight loss
Maternal satisfaction with postpartum care assessed through surveys/interviews | 3, 6, and 12 months postpartum
  Assessment of maternal satisfaction with postpartum care elicited through self-administered surveys and/or provider interviews.
Identification of a primary care provider elicited through interviews | 3, 6, and 12 months postpartum
  Identification of a primary care provider elicited through interviews with providers

CONTACTS AND LOCATIONS:
Overall Officials: Jenifer Fahey, CNM, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No